CLINICAL TRIAL: NCT02613676
Title: Transcutaneous Screening for Risk of Severe Hyperbilirubinemia in South African Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Charles Okwundu, Researcher, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: TcBScreening
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Neonatal Jaundice; Hyperbilirubinemia
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia | interventions — Standard of Care; Watchful Waiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TcB screening before discharge (Experimental): Participants in this group will be screened for jaundice using the JM 105 transcutaneous device. The TcB value will be plotted on the Bhutani nomogram to assess the risk category. Infants who are categorised as high risk according to the nomogram will require blood sampling for TsB and assessment for need for phototherapy.
  Interventions: Device: Transcutaneous bilirubin screening
- Standard care (visual inspection) (Other): Participants in this group will be managed routinely according to the current standard of care where babies are assessed for jaundice by visual inspection. Babies in this group will require blood draw for TsB if there are visibly jaundiced
  Interventions: Other: Standard care (Visual inspection)

INTERVENTIONS:
Device: Transcutaneous bilirubin screening — Transcutaneous bilirubin screening before hospital discharge and assessment of risk category according to the Bhutani nomogram
  Arms: TcB screening before discharge
Other: Standard care (Visual inspection) — Participants in this group will be assessed for jaundice by visual inspection. Blood draw for TsB will be drawn only if the participant is visibly jaundiced.
  Arms: Standard care (visual inspection)

SUMMARY:
In South Africa, healthy term newborns are usually discharged early (<72 hours after delivery). Many studies have shown that hospital readmission rates have increased with this practice, and jaundice or hyperbilirubinemia is the most common cause of readmission of newborns. Peak serum bilirubin levels usually occur on postnatal days 3-5, by when many have already been discharged putting the infant at increased risk of severe hyperbilirubinemia. Severe neonatal jaundice still constitutes an important cause of neonatal mortality and morbidity in Africa. Screening all newborns for the risk of severe hyperbilirubinemia before hospital could help in early identification of hyperbilirubinemia and early intervention and potentially prevent unwanted consequences like bilirubin induced neurological dysfunction. However, there are conflicting recommendations on the use of universal transcutaneous bilirubin screening for jaundice in all newborns before hospital discharge.

DETAILED DESCRIPTION:
Like in many other countries in Africa and the rest of the world, objective screening for risk of severe hyperbilirubinemia using serum bilirubin (TsB) or transcutaneous bilirubin (TcB) measurement is currently not standard of care in South Africa. The investigators therefore propose to test the use of a non-invasive TcB device to detect and predict the risk of severe jaundice before discharge of babies from the new-born nursery in a South African population of newborns.

OBJECTIVE To evaluate the effects of transcutaneous bilirubin screening in newborns before hospital discharge.

METHODS In this randomised controlled trial (RCT) the investigators will compare the traditional visual assessment and TcB measurement before hospital discharge. About 1858 newborns ≥35 weeks gestational age and/or ≥1800 g, who are <72 hrs of life will be randomly allocated into two groups: a) TcB screening, or b) visual assessment (standard care)

Subjects:

Babies ≥ 35 wks gestational age and/or ≥ 1800g, who are <72 hrs of life.

Study arms:

Participants will be randomised within 72 hrs of birth into: a) TcB screening plotted on the nomogram or b) visual assessment of jaundice.

Control group (Standard care):

In this group, participants will be assessed for jaundice by the use of the traditional visual assessment before discharge. A formal serum bilirubin level will be done on all infants who are visibly jaundiced and decide on need for phototherapy.

TcB screening group:

All participants in this group, will be assessed for the risk of severe hyperbilirubinemia by measurement of bilirubin level using the JM 105 transcutaneous device at < 72 hrs of life before hospital discharge. The bilirubin level will be plotted on the Bhutani hour-specific nomogram to determine the risk zone. Babies will be classified into four different different risk categories: high-risk, high-intermediate, low-intermediate and low risk categories depending on the transcutaneous bilirubin level. Follow-up or intervention will be planned based on the risk category. For participants who are identified as high risk for severe hyperbilirubinemia, the investigators will perform a formal TsB measurement and determine need for phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* All newborns ≥ 35 wks gestational age and ≥ 1800g
* Babies who who are < 72 hours of life

Exclusion Criteria:

* Prior use of phototherapy
* Major congenital anomaly
* Babies born < 35 wks gestational age or < 1800g

Ages: 6 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1858 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Readmission for hyperbilirubinemia | Up to two weeks
  The primary outcome is readmission for hyperbilirubinemia requiring phototherapy or exchange transfusion

SECONDARY OUTCOMES:
Phototherapy before discharge | Up to two weeks
  This outcome refers to the use of phototherapy for the treatment of hyperbilirubinemia before hospital discharge.
TsB > 427 umol/l or TsB > threshold for exchange transfusion | Up to two weeks
Length of hospital stay (days) | Up to two weeks
Blood draw for total serum bilirubin | Up to two week
  This outcome refers to blood sampling for laboratory measurement of TsB

CONTACTS AND LOCATIONS:
Overall Officials: Charles I Okwundu, MBBS, MPH, Principal Investigator — University of Stellenbosch; Vinod K Bhutani, MD, Principal Investigator — Stanford University
Locations (1):
- Tygerberg Hospital, Cape Town, Western Cape, South Africa